CLINICAL TRIAL: NCT05760235
Title: Prospective Pilot Study for the Evaluation of Endoscopic Sleeve Gastroplasty With Endomina® for the Treatment of Obesity in Liver Transplant Candidates
Acronym: ESGiTX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4903
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Liver Transplantation; Obesity; Bariatric Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver transplant obese candidates (Experimental): Subjects with an indication to liver transplantation that are not listed because of a high BMI according to the policy of the transplant Centre (cut-off 35 kg/m2)
  Interventions: Procedure: Endoscopic sleeve gastroplasty (ESG)

INTERVENTIONS:
Procedure: Endoscopic sleeve gastroplasty (ESG) — ESG will be performed under general anaesthesia with orotracheal intubation. The Endomina® suturing system (EndoTools Therapeutics S.A., Gosselies, Belgium) mounted on a single channel endoscope will be used. This system allows to obtain full thickness gastric sutures through the gastric wall of the gastric body, leaving the antrum and the gastric fundus free15. The procedure will be performed with the patient in supine position. Carbon dioxide will be blown to stretch the gastric lumen. An initial endoscopic evaluation will be performed immediately to confirm the absence of any contraindication to ESG before suturing. The ESG starts with the reduction of the gastric body, suturing from distal to proximal and starting from the notch of the angulus and ending at the level of the fundus. 4-8 full thickness stitches will be placed, with 2 passes per stitch.

SUMMARY:
The goal of this pilot prospective interventional study is to evaluate the efficacy of endoscopic sleeve gastroplasty (ESG) in allowing obese subjects with the need of liver transplantation to reduce their BMI in order to enter the waiting list (BMI (≥35 kg/m2). The main question[s] it aims to answer are:

* Is the procedure effective in reducing BMI to the target level in 12 months?
* Which is the effect on weight loss, quality of life and obesity-related comorbidities?

Participants will undergo ESG as per standard clinical practice and followed up to 12 months before transplantation and for 12 months after transplantation

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (i.e., age between 18 and 70 years).
* BMI ≥ 35 kg/m²;
* Subjects with an indication to liver transplantation that are not listed because of a high BMI according to the policy of the transplant Centre (cut-off 35 kg/m2);
* Signed informed consent.

Exclusion Criteria:

* Clinically significant portal hypertension at upper endoscopy: F3 or F1/F2 with red signs oesophageal varices, gastric varices or severe hypertensive gastropathy;
* Upper gastro-intestinal bleeding (gastric or esophageal) in the previous six months;
* CHILD C class;
* Clinically or ultrasound-detected ascites in the 15 days before the procedure. Only mild ascitic effusion in the pelvis will be accepted;
* Spontaneous bacterial peritonitis in the previous 6 months;
* Hepatocellular carcinoma with extra hepatic spread;
* Previous stomach, oesophagus or duodenum surgery;
* Technical non-feasibility in the opinion of the endoscopist;
* Clinical signs of active infection;
* Unstable cardiac disease or chronic heart failure;
* Platelet count less than 70.000;
* International Normalized Ratio ≥ 1,5;
* Concomitant unstoppable anticoagulant or anti platelet therapy, except for low dose aspirin (≤ 100 mg);
* Acute liver failure;
* Easy to bleed during diagnostic endoscopy;
* Active drugs or alcohol abuse;
* Pregnancy, lactation (desire to become pregnant during study duration);
* Enrolment in other clinical studies;
* Contraindication to general anaesthesia;
* Contraindication to endoscopic procedure;
* Other conditions to exclude the subject in investigators opinion;
* Refusal to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Transplant list inclusion | 12 months
  number of patients who achieve a BMI < 35 kg/m² within 12 months post-ESG, allowing them to be included in the transplant list

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Lazio, Italy